CLINICAL TRIAL: NCT04052451
Title: The Safety, Efficacy, and Tolerability of Microbial Ecosystem Therapeutic-2 in People With Major Depression and/or Generalized Anxiety Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NuBiyota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MET-2-301
Record Dates: First submitted 2019-08-08; First posted 2019-08-09 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2019-08

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This is an open label study with one arm for subjects diagnosed with major depression disorder and one arm for subjects diagnosed with generalized anxiety disorder
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Major Depression Disorder (Experimental): MET-2 will be given to subjects with major depression disorder and its effect on mood will be measured
  Interventions: Biological: MET-2
- Generalized Anxiety Disorder (Experimental): MET-2 will be given to subjects with generalized anxiety disorder and its effect on mood will be measured
  Interventions: Biological: MET-2

INTERVENTIONS:
Biological: MET-2 — Subjects will take study medication once daily for the duration of the study

SUMMARY:
This study will measure the effects of MET-2 on symptoms of depression and anxiety using pre- and post-treatment scores for overall depression and anxiety and other symptoms of depression, such as sleep and anhedonia.

DETAILED DESCRIPTION:
This study will measure the effects of MET-2 on symptoms of depression and anxiety using pre- and post-treatment scores for overall depression and anxiety and other symptoms of depression, such as sleep and anhedonia.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent.
2. Not pregnant
3. Willing to participate in follow up as part of the study
4. Diagnosis of MDD and/or GAD by MINI
5. Current depressive episode with a MADRS score of ≥15 or Current GAD episode with GAD-7 score of ≥8.
6. Able to understand and comply with the requirements of the study
7. Able to provide stool and blood samples.

Exclusion Criteria:

1. History of chronic diarrhea
2. Need for regular use of agents that affect GI motility (narcotics such as codeine or morphine, agents such as loperamide or metoclopramide)
3. Colostomy
4. Elective surgery that will require preoperative antibiotics planned within 6 months of enrolment
5. Pregnant, breastfeeding, or planning to get pregnant in the next 6 months
6. Any condition for which, in the opinion of the investigator, the participant should be excluded from the study.
7. Current use of any antidepressant/antianxiety drug (eligible to participate after a 4-week washout period)
8. Use of any antibiotic drug in the past 4 weeks (may be eligible to participate after a 1-month washout period)
9. History of alcohol or substance dependence in the past 6 months
10. Daily use of probiotic product in the past 2 weeks (may be eligible to participate after a 2-week washout period)
11. Use of any type of laxative in the last 2 weeks.
12. Consumption of products fortified in probiotics
13. High suicidal risk, as measured by MADRS item 10 score more than 3 (or 4)
14. Current psychotic symptoms
15. Bipolar Depression
16. History of epilepsy or uncontrolled seizures
17. Immunodeficiency (immuno-compromised and immuno-suppressed participants; e.g. acquired immune deficiency syndrome [AIDS], lymphoma, participants undergoing long-term corticosteroid treatment, chemotherapy and allograft participants)
18. Unstable medical conditions or serious diseases/conditions (e.g. cancer, cardiovascular, renal, lung, diabetes, psychiatric illness, bleeding disorders, etc.)
19. The use of natural health products (Natural health products [NHPs]; e.g. St. John's Wort, passion flower, etc.) that affect depression
20. History of Electroconvulsive therapy (ECT)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | Week 10
  The MADRS is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders
Generalized Anxiety Disorder - 7 (GAD-7) | Week 10
  The GAD-7 is a seven domain, self-reported questionnaire for screening and assessing severity of generalized anxiety disorder.

CONTACTS AND LOCATIONS:
Locations (1):
- Providence Care Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Derived] Chinna Meyyappan A, Forth E, Milev R. Microbial Ecosystem Therapeutic-2 Intervention in People With Major Depressive Disorder and Generalized Anxiety Disorder: Phase 1, Open-Label Study. Interact J Med Res. 2022 Jan 21;11(1):e32234. doi: 10.2196/32234. PMID 35060914